CLINICAL TRIAL: NCT01064544
Title: Effects of Light Therapy on Sleep, Melatonin Rhythm and Mood in Hemodialysis Patients
Brief Title: Study on Hemodialysis: Illumination Effects
Acronym: SHINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meander Medical Center (Other)
Responsible Party: Department of Clinical Pharmacy, Meande Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R-09.37 M / SHINE
Record Dates: First submitted 2010-02-03; First posted 2010-02-08 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Sleep Problems
Keywords: Sleep problems; melatonin; mood; Hemodialysis
MeSH Terms: conditions — Parasomnias | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Starting with light therapy (Experimental): Starts with 3 weeks of light therapy, followed by a control period
  Interventions: Procedure: light therapy with the device: EnergyLight
- Ending with light therapy (Experimental): Ends with 3 weeks of light therapy after a control period.
  Interventions: Procedure: light therapy with the device: EnergyLight

INTERVENTIONS:
Procedure: light therapy with the device: EnergyLight — 2 hr of light therapy during each hemodialysis session
  Other Names: Philips Energylight

SUMMARY:
Previous research has shown that sleep quality in hemodialysis patients is disturbed. One of the possible explanations is an insufficient or disturbed melatonin rhythm. Melatonin rhythm is regulated by exposure to light. In this feasibility study, the investigators examine the effects of light therapy during dialysis on sleep, melatonin rhythm and mood.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* men/women aged 18-85 years
* knowledge of the dutch language
* hemodialysis patient
* subjective sleep problems (Epworth sleepiness score >9)

Exclusion Criteria:

* known major illness, which interferes with patient's participation
* use of melatonin/hypnotics
* use of photosensitizing medication
* jet lag or travel > 1 time zone

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Improvement of sleep parameters | 3 weeks

SECONDARY OUTCOMES:
Change in subjective sleep parameters | 3 weeks
Change in mood | 3 weeks
change in melatonin concentrations | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gaillard, MD, PhD, Study Chair — Meander Medical Center
Locations (1):
- Meander Medical Center, Amersfoort, Netherlands